CLINICAL TRIAL: NCT05646368
Title: A Randomized, Crossover Study to Assess Bioavailability of Select Nutrients From Two Formulations of a Multivitamin/Mineral Supplement in Healthy Adults
Brief Title: Bioavailability of Select Nutrients From Two Formulations of a Multivitamin/Mineral Supplement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Midwest Center for Metabolic and Cardiovascular Research (Other)
Collaborators: Pharmavite LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: MB-2113
Record Dates: First submitted 2022-12-01; First posted 2022-12-12 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Bioavailability
MeSH Terms: interventions — Akacid-medical-formulation

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Formulation #1 of a multivitamin/mineral supplement (Experimental): Subject will receive a single dose of formulation #1 of a multivitamin/mineral supplement
  Interventions: Dietary Supplement: Formulation #1
- Formulation #2 of a multivitamin/mineral supplement (Active Comparator): Subject will receive a single dose of formulation #2 of a multivitamin/mineral supplement
  Interventions: Dietary Supplement: Formulation #2

INTERVENTIONS:
Dietary Supplement: Formulation #1 — Subject will receive a single dose of formulation #1 of a multivitamin/mineral supplement
  Arms: Formulation #1 of a multivitamin/mineral supplement
Dietary Supplement: Formulation #2 — Subject will receive a single dose of formulation #2 of a multivitamin/mineral supplement
  Arms: Formulation #2 of a multivitamin/mineral supplement

SUMMARY:
The objective of this study is to assess the relative bioavailability of select nutrients from two formulations of a multivitamin/mineral supplement in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male or female, 18 to 45 years of age, inclusive.
2. Subject has a BMI of ≥18.50 and <30.00 kg/m2.
3. Subject is a non-smoker (at least 6 months) and has no plans to start smoking (or vaping) during the study period.
4. Subject is judged to be in good health based on medical history and routine laboratory tests.
5. Subject has a score of ≥7 on the Vein Access Scale.
6. Subject agrees to abstain from alcohol consumption and vigorous physical activity for at least 24 h prior to all test visits.
7. Subject understands the study procedures, and is willing to complete them, and signs forms documenting informed consent to participate in the study and authorization for release of relevant protected health information to the study Investigator.

Exclusion Criteria:

1. Individual has a history of difficulty swallowing capsules or large pills.
2. Individual has a serum folate concentration outside of the normal range (>3.0 ng/ml) at visit 1, day -7.
3. Individual has a serum zinc concentration outside of the normal range (44-115 μg/dL) on visit 1, day -7.
4. Individual has a serum magnesium concentration outside of the normal range (1.6 - 2.3 mg/dL) on visit 1, day -7.
5. Individual has a serum vitamin B12 concentration outside of the normal range (232-1245 pg/mL) on visit 1, day -7.
6. Individual has a hemoglobin outside of the normal range (13.0-17.7 g/dL).
7. Individual has had a blood transfusion during the 3 months prior to the screening visit (visit 1, day -7).
8. Individual has any gastrointestinal condition that would potentially interfere with absorption of the study product (e.g., inflammatory bowel disease, celiac disease, history of gastric bypass surgery, chronic gastritis).
9. Individual has a history or presence of clinically important medical diagnosis, in the opinion of the Principal Investigator.
10. Individual has an active infection or sign/symptoms of an infection. The test days (visits 2-5) will be rescheduled to allow the subject to be symptom-free of any type of systemic infection for at least five days.
11. Individual has recent use of antibiotics (within 7 days of visit 2, day 0) and throughout the study period. The test days will be rescheduled to allow the subject to wash out the antibiotic for at least 7 days.
12. Individual has unstable use (initiation or change in dose) within four weeks of visit 2 (day 0) of antihypertensive medications, thyroid hormone replacement, hormonal contraceptives, or hormone therapy.
13. Individual has consumed any dietary supplements (including all vitamin/mineral supplements) within one week of visit 2, day 0 and throughout the study period.
14. Individual has received an intramuscular injection of vitamin B12 within 6 months of visit 2, day 0.
15. Subject is female who is pregnant, planning to be pregnant during the study period, lactating, or is of childbearing potential and is unwilling to commit to the use of a medically approved form of contraception throughout the study period.
16. Individual has consumed alcoholic beverages within 24 h of each test day visit (visits 2-5).
17. Individual has used medications known to interfere with vitamin and mineral absorption within one week of visit 2, day 0 and throughout the study period, including but not limited to, aspirin, anti-inflammatories, antacids, histamine 2 receptor antagonists, and proton-pump inhibitors.
18. Individual is taking an anticonvulsant medication.
19. Individual has extreme dietary habits, as judged by the Investigator (e.g., vegan, Atkins, very low carbohydrate/very high protein, etc.).
20. Individual has history of an eating disorder (e.g., anorexia nervosa, bulimia nervosa, binge eating) diagnosed by a health professional.
21. Individual has any major trauma or surgical event within 12 weeks of the screening visit (visit 1, day -7).
22. Individual has uncontrolled hypertension (systolic blood pressure ≥160 mm Hg and/or diastolic blood pressure ≥100 mm Hg) at screening (visit 1, day -7). One re-test will be allowed on a separate day prior to visit 2, day 0 for subjects whose blood pressure exceeds either of these cut points at visit 1.
23. Individual has a recent history or strong potential for drug or alcohol abuse or has a positive urine drug screen.
24. Individual has a known allergy to any ingredients in the study products or provided meals/snacks.
25. Individual has a condition the Investigator believes would interfere with her ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results or put the person at undue risk.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-12-23 (Actual); Primary Completion 2023-05-04 (Actual); Study Completion 2023-05-04 (Actual)

PRIMARY OUTCOMES:
Baseline-adjusted geometric mean ratio (GMR) for area under the curve (AUC) from 0 to 2 h for plasma folate | Baseline to 2 hours
  Changes in GMR for baseline-adjusted AUC for plasma folate

SECONDARY OUTCOMES:
Unadjusted and baseline-adjusted AUC from 0 to 2 h for select nutrients in plasma | Baseline to 2 hours
  Changes in unadjusted and baseline-adjusted AUC for select nutrients in plasma
Unadjusted and baseline-adjusted GMRs for AUC from 0 to 2 h for select nutrients in plasma | Baseline to 2 hours
  Changes in unadjusted and baseline-adjusted GMRs for AUC for select nutrients in plasma
Unadjusted and baseline-adjusted AUC from 0 to 8 h for select nutrients in plasma | Baseline to 8 hours
  Changes in unadjusted and baseline-adjusted AUC for select nutrients in plasma
Unadjusted and baseline-adjusted GMRs for AUC from 0 to 8 h for select nutrients in plasma | Baseline to 8 hours
  Changes in unadjusted and baseline-adjusted GMRs for AUC for select nutrients in plasma
Maximum concentrations of select nutrients in plasma | Baseline to 8 hours
  Differences between study products in unadjusted and baseline-adjusted maximum concentrations of select nutrients in plasma
Time (in hours) to reach the maximum concentration of select nutrients in plasma | Baseline to 8 hours
  Differences between study products in the time to reach the maximum concentration of select nutrients in plasma
Concentration of a select nutrient in urine | Baseline to 24 hours
  Differences between study products in the concentration of a select nutrient in urine

CONTACTS AND LOCATIONS:
Overall Officials: Kevin C Maki, PhD, Study Director — MB Clinical Research & Consulting
Locations (1):
- Health Awareness, Port Saint Lucie, Florida, United States

IPD SHARING:
Plan to Share IPD: No